CLINICAL TRIAL: NCT01844791
Title: A Phase IIa Exploratory Study of OCZ103-OS in Combination With Platinum-Gemcitabine Based Doublet First Line Therapy in Stage IV Non-Small Cell Lung Cancer (NSCLC) Patients
Brief Title: An Exploratory Study of OCZ103-OS in Combination With Standard of Care in Stage IV Non-Small Cell Lung Cancer (NSCLC) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncozyme Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCZ103-206
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; OCZ103-OS; Pentamidine bis(2-hydroxyethanesulfonate); platinum-gemcitabine based doublet first line therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Platinum; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OCZ103-OS, Platinum, Gemcitabine (Experimental): OCZ103-OS in combination with Platinum-Gemcitabine as standard of care
  Interventions: Drug: OCZ103-OS; Drug: Platinum; Drug: Gemcitabine

INTERVENTIONS:
Drug: OCZ103-OS — OCZ103-OS is given in combination with chemotherapy each cycle
  Other Names: pentamidine bis(2-hydroxyethanesulfonate
Drug: Platinum — Platinum is given as standard chemotherapy each cycle
Drug: Gemcitabine — Gemcitabine is given as standard chemotherapy each cycle

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of the use of OCZ103-OS in combination with Platinum-Gemcitabine based doublet first line therapy in stage IV non-small cell lung cancer (NSCLC) patients.

DETAILED DESCRIPTION:
This is a single arm, open label study to investigate the safety and efficacy of the use of OCZ103-OS in combination with Platinum-gemcitabine base doublet first line therapy in stage IV non-small cell lung cancer (NSCLC) patients.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent;
* Males or females;
* 18-75 years;
* Histologically or cytologically confirmed stage IV NSCLC patients that are eligible to platinum-gemcitabine based doublet therapy (M1a and M1b, seventh edition descriptor of the Revised International System for Staging Lung Cancer, adopted by the AJCC.) Patients with a prior diagnosis of stage IIIa or IIIb NSCLC who have progressed to stage IV are also eligible;
* ECOG performance 0 or 1;
* One or more tumor lesions measurable by RECIST criteria version 1.1, on CT scan or MRI;
* Patients with previous radiotherapy as definitive therapy for locally advanced non-small cell lung cancer are eligible, as long as the selected measurable lesions are outside the original radiation therapy port unless there has been demonstrated progression in the lesion. Radiation therapy must have been completed > 4 weeks prior to study entry;
* Palliative radiotherapy must have been completed > 2 weeks prior to study entry. Concomitant palliative radiotherapy to an existing bone lesion for pain control is allowed;
* Life expectancy of at least 3 months

Exclusion Criteria:

* Any prior systemic therapy for recurrent or metastatic NSCLC, except prior neoadjuvant or adjuvant systemic chemotherapy for NSCLC if administered at least 6 months prior to enrolment;
* Any of the following conditions: Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥ 2; atrial fibrillation of any grade; QTc interval > 450 msec for males or > 470 msec for females or uncontrolled intercurrent illness, e.g. unstable angina; severe coronary disease, ventricular arrhythmias, bradycardia < 50 bpm; a history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia or family history of Long QT Syndrome);
* Systolic Blood Pressure < 100 mmHg (if deemed clinically significant by the treating physician);
* Uncontrolled diabetes. Patients with well controlled diabetes, with a HbA1C of less than 7%, on stable hypoglycaemic therapy and diet, are eligible;
* Clinically significant renal impairment or chronic pancreatitis;
* History of clinically significant hypoglycemia, with fasting blood glucose < 3 mmol/L;
* Inadequate baseline organ function as shown by following laboratory values:
* Hemoglobin < 100 g/L
* Absolute neutrophil count <1.5 x 10e9/L
* Platelet count < 100 x 10e9/L
* Total bilirubin > 1.5 x ULN
* AST and ALT > 2.5 x ULN or > 5 ULN in the presence of liver metastases
* Serum creatinine > 1.5 x ULN or calculated creatinine clearance < 60 ml/min
* To be dependent of oxygen treatment;
* Active infections requiring antibiotics;
* A major surgical procedure, open biopsy, or significant traumatic injury within 28 days of beginning treatment, or anticipation of the need for major surgery during the course of the study;
* Pregnancy or breastfeeding. All women of child-bearing potential must have a negative pregnancy test prior to first receiving protocol therapy;
* Active alcohol or drug abuse;
* Known or suspected allergy/hypersensitivity to any agent given in the course of this trial;
* Any co-morbid condition that in the judgment of the investigator renders the subject at high risk of treatment complication or reduces the probability of assessing clinical effect;
* Other malignancies diagnosed within the last 5 years with the exception of Basal Cell Carcinoma of the skin;
* Patients unable to comply with the study protocol and follow-up schedule for any psychological, familial, sociological or geographical reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Overall Response | one year four months
  To assess the effect of OCZ103-OS on overall objective response in subjects with stage IV non-small cell lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Kalinka-Warzocha, MD-PhD, Study Director — Wojewodzki Szpital Specjalistyczny im .M. Kopernika w
Locations (1):
- Ewa Kalinka-Warzocha, Lodz, Poland